CLINICAL TRIAL: NCT02979691
Title: A Phase II/III Study Comparing Simultaneous Integrated Boost (SIB) Intensity Modulated Radiation Therapy (IMRT) With S1 Based SIB-IMRT Followed by Adjuvant Chemotherapy With S1 in Elderly Patients With Esophageal or Esophagogastric Cancer (3JECROG-P01)
Brief Title: Phase II/III Study Comparing Chemoradiotherapy With Radiotherapy in Elderly Patients With Esophageal or Esophagogastric Cancer - 3JECROG P-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Anyang Tumor Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Affiliated Hospital of Hebei University (Other); Fujian Cancer Hospital (Other Government); Tengzhou Central People's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Dr., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3JECROG P-01
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Esophagus Cancer; Esophagogastric Junction Cancer; Radiotherapy; Complications; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination)

ARMS (2):
- SIB-IMRT (Active Comparator): SIB-IMRT arm receives intensity-modulated radiotherapy with a simultaneous integrated boost (SIB-IMRT) (59.92Gy and 50.4Gy in 28 fractions) concurrently with oral S-1(40-60mg, orally twice daily, on every weekday).
  Interventions: Radiation: SIB-IMRT
- S1 based SIB-IMRT (Experimental): S1 based SIB-IMRT receives intensity-modulated radiotherapy with a simultaneous integrated boost (SIB-IMRT) (59.92Gy and 50.4Gy in 28 fractions) concurrently with oral S-1(40-60mg, orally twice daily, on every weekday) followed by four cycles of S-1 (40-60mg, orally twice daily, d1-14, every 3 weeks) as an adjuvant chemotherapy.
  Interventions: Radiation: SIB-IMRT; Drug: S-1

INTERVENTIONS:
Radiation: SIB-IMRT
Drug: S-1
  Arms: S1 based SIB-IMRT

SUMMARY:
Ratiotherapy alone is the current standard treatment for elderly esophageal or esophagogastric cancer in China. And Little is known about chemoradiotherapy (CRT) in elderly patients. This study aimed to assess the efficiency and safety of simultaneous integrated boost (SIB) intensity modulated radiation therapy (IMRT) with S1 based SIB-IMRT followed by adjuvant chemotherapy with S1 in in elderly (age ≥70 years) esophageal or esophagogastric cancer patients

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years
* Esophageal or Esophagogastric cancer
* Histologically proven squamous cell carcinoma or adenocarcinoma in patients staged as IIa-IVb (UICC 2002, IVb only with supraclavicular or celiac trunk lymph nodes metastasis)
* Karnofsky performance status(KPS)≥ 70 and Charlson score ≤3
* No distant metastasis other than supraclavicular lymph nodes
* No prior history of thoracic radiation
* Patients must have normal organ and marrow function as defined below: Leukocytes: greater than or equal to 3,500 G/L; Platelets: greater than or equal to 100,000/mm3 .Hemoglobin:greater than or equal to 10g/L .Total bilirubin: within normal institutional limits; AST/ALT: less than or equal to 1.5 times the upper limit; Creatinine within normal upper limits
* Informed consent

Exclusion Criteria:

* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* With any distant metastasis out of regional lymphatic drainage or in liver,lung,bone,CNS,etc
* History of allergic reactions attributed to similar chemical or biologic complex to S-1
* With esophageal fistula, perforation, cachexia prior to treatment
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* Pregnant or lactating females

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Comprehensive geriatric assessment | Baseline
  A comprehensive geriatric assessment (CGA) is a multidisciplinary evaluation in which multiple problems of older persons are described.It consists several questionnaires used to assess an older individual's functional status,comorbid medical condition,cognition, psychologic state, social support, and nutritional status,etc.
Remission rate of dysphagia | Change from baseline to 1 month after treatment
Progression free survival | 1 year
Time of locoregional control and failure site within or outside radiation field | 1 year
Radiotherapy toxicities | 2 months
Chemoradiotherapy toxicities | 2 months

OTHER OUTCOMES:
Analysis of relationship between dosimetric parameters of radiation technique and acute or late side effects | 6 months
CT/MRI Texture Features in evaluating the tumor response and prognosis | Change from baseline to 1 month after treatment
Clinical target contouring guided by MRI or CT simulation | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Derived] Wang X, Han W, Zhang W, Wang X, Ge X, Lin Y, Zhou H, Hu M, Wang W, Liu K, Lu J, Qie S, Zhang J, Deng W, Wang L, Han C, Li M, Zhang K, Li L, Wang Q, Shi H, Yu Z, Zhao Y, Sun X, Shi Y, Pang Q, Zhou Z, Liang J, Chen D, Feng Q, Bi N, Zhang T, Deng L, Wang W, Liu W, Wang J, Zhai Y, Wang J, Chen W, Chen J, Xiao Z; Jing-Jin-Ji Esophageal and Esophagogastric Cancer Radiotherapy Oncology Group (3JECROG). Effectiveness of S-1-Based Chemoradiotherapy in Patients 70 Years and Older With Esophageal Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312625. doi: 10.1001/jamanetworkopen.2023.12625. PMID 37195667
- [Derived] Wang X, Ge X, Wang X, Zhang W, Zhou H, Lin Y, Qie S, Hu M, Wang W, Liu K, Pang Q, Li M, Chen J, Liu M, Zhang K, Li L, Shi Y, Deng W, Li C, Ni W, Chang X, Han W, Deng L, Wang W, Liang J, Bi N, Zhang T, Liu W, Wang J, Zhai Y, Feng Q, Chen D, Zhou Z, Zhao Y, Sun X, Xiao Z. S-1-Based Chemoradiotherapy Followed by Consolidation Chemotherapy With S-1 in Elderly Patients With Esophageal Squamous Cell Carcinoma: A Multicenter Phase II Trial. Front Oncol. 2020 Aug 28;10:1499. doi: 10.3389/fonc.2020.01499. eCollection 2020. PMID 32983991
- [Derived] Li C, Wang X, Wang X, Han C, Wang P, Pang Q, Chen J, Sun X, Wang L, Zhang W, Lin Y, Ge X, Zhou Z, Ni W, Chang X, Liang J, Deng L, Wang W, Zhao Y, Xiao Z. A multicenter phase III study comparing Simultaneous Integrated Boost (SIB) radiotherapy concurrent and consolidated with S-1 versus SIB alone in elderly patients with esophageal and esophagogastric cancer - the 3JECROG P-01 study protocol. BMC Cancer. 2019 Apr 29;19(1):397. doi: 10.1186/s12885-019-5544-1. PMID 31036088